CLINICAL TRIAL: NCT06211036
Title: A Phase 3, Open-label, Multicenter, Randomized Study of Tarlatamab in Combination With Durvalumab vs Durvalumab Alone in Subjects With Extensive-Stage Small-Cell Lung Cancer Following Platinum, Etoposide and Durvalumab (DeLLphi-305)
Brief Title: Study Comparing Tarlatamab and Durvalumab Versus Durvalumab Alone in First-Line Extensive-Stage Small-Cell Lung Cancer (ES-SCLC) Following Platinum, Etoposide and Durvalumab
Acronym: DeLLphi-305
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200041; 2023-505989-29 (Other: EU CT Number)
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Extensive-Stage Small-Cell Lung Cancer; Small-Cell Lung Cancer
Keywords: Extensive-Stage Small-Cell Lung Cancer; ES-SCLC; Platinum; Etoposide; Durvalumab; Tarlatamab; AMG 757
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — AMG 757; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tarlatamab in Combination With Durvalumab (Experimental): Participants will receive tarlatamab once every 2 weeks (Q2W) and durvalumab once every 4 weeks (Q4W).
  Interventions: Drug: Tarlatamab; Drug: Durvalumab
- Durvalumab Alone (Active Comparator): Participants will receive durvalumab Q4W alone.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Tarlatamab — Intravenous (IV) infusion
  Other Names: AMG 757
  Arms: Tarlatamab in Combination With Durvalumab
Drug: Durvalumab — IV infusion

SUMMARY:
The primary objective of this study is to compare the efficacy of tarlatamab plus durvalumab with durvalumab alone on prolonging overall survival (OS).

ELIGIBILITY:
Inclusion:

* Participant has provided informed consent prior to initiation of any study specific activities/procedures.
* Age >= 18 years (or >= legal adult age within the country if it is older than 18 years).
* Completed 3-4 cycles of platinum-etoposide chemotherapy with concurrent durvalumab as first-line treatment of extensive-stage (ES)-SCLC prior to enrollment, without disease progression (ongoing response or stable disease) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 1.
* Minimum life expectancy > 12 weeks.
* Toxicities attributed to prior anti-cancer therapy resolved to grade ≤ 1, unless otherwise specified, excluding alopecia or fatigue.
* Adequate organ function.
* Histologically or cytologically documented extensive-stage disease (American Joint Committee on Cancer, 2017, IV small-cell lung cancer (SCLC) [T any, N any, M1 a/b/c]), or T3 to T4 due to multiple lung nodules that are too extensive or have tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan. Participants with prior limited-stage (LS)-SCLC are allowed if the interval is > 6 months since the end of previous therapy and progression, in discussion with the medical monitor.

Exclusion

* Symptomatic central nervous system (CNS) metastases, or leptomeningeal disease. Participants with treated brain metastases are eligible as per protocol.
* Prior history of severe or life-threatening events from any immune-mediated therapy.
* History of other malignancy within the past 2 years, with some exceptions as per protocol.
* Active or prior documented autoimmune or inflammatory disorders as per protocol.
* Myocardial infarction and/or symptomatic congestive heart failure (New York Heart Association > class II) within 6 months of first dose of study treatment.
* History of arterial thrombosis (e.g., stroke or transient ischemic attack) within 6 months of first dose of study treatment.
* Evidence of interstitial lung disease (ILD) or active, non-infectious pneumonitis.
* History of solid organ transplant.
* Major surgical procedures within 28 days of first dose of study treatment.
* Known human immunodeficiency virus (HIV) infection (participants with HIV infection on antiviral therapy and undetectable viral load are permitted with a requirement for regular monitoring for reactivation for the duration of treatment on study), hepatitis C infection (participants with hepatitis C that achieve a sustained virologic response after antiviral therapy are allowed), or hepatitis B infection (participants with hepatitis B surface antigen [HBsAg] or core antibody that achieve sustained virologic response with antiviral therapy are permitted with a requirement for regular monitoring for reactivation for the duration of treatment on the study).
* Receiving systemic corticosteroid therapy or any other form of immunosuppressive therapy within 14 days prior to first dose of study treatment.
* History of allergic reactions or acute hypersensitivity reaction to antibody therapies, platinum chemotherapy, or etoposide.
* Participant with symptoms and/or clinical signs and/or radiographic signs that indicate an acute and/or uncontrolled active systemic infection within 7 days prior to the first dose of study treatment.
* Participant has known active infection requiring parenteral antibiotic treatment. Upon completion of parenteral antibiotics and resolution of symptoms, the participant may be considered eligible for the study from an infection standpoint.
* Treatment with live virus, including live-attenuated vaccination, within 4 weeks prior to the first dose of study treatment. Inactive vaccines (e.g., non-live or non-replicating agent) and live viral non-replicating vaccines (e.g., Jynneos for Monkeypox infection) within 30 days prior to first dose of study treatment.
* Prior therapy with any selective inhibitor of the delta-like ligand 3 (DLL3) pathway.
* Receiving another anti-cancer therapy. Adjuvant hormonal therapy for resected breast cancer is permitted.
* Treatment in an alternative investigational trial within 28 days prior to enrollment.
* Has received or is planning to receive consolidative chest radiation for extensive stage disease.
* Female participants of childbearing potential unwilling to use protocol specified method of contraception during treatment as per protocol.
* Female participants who are breastfeeding or who plan to breastfeed while on study as per protocol.
* Female participants planning to become pregnant or donate eggs while on study as per protocol.
* Female participants of childbearing potential with a positive pregnancy test assessed at screening by a highly sensitive serum pregnancy test.
* Male participants with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception during treatment as per protocol.
* Male participants with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment as per protocol.
* Male participants unwilling to abstain from donating sperm during treatment as per protocol.
* Participant has known sensitivity to any of the products or components to be administered during dosing.
* Participant has known sensitivity to any of the products or components to be administered during dosing.
* History or evidence of any other clinically significant disorder, condition or disease that, in the opinion of the investigator or physician if consulted, would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.
* Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (eg, Clinical Outcome Assessments) to the best of the participant and investigator's knowledge. Participants who are unable to complete clinical outcome assessments are eligible.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 563 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2027-07-05 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
OS | Up to approximately 3 years

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 3 years
Overall Response (OR) | Up to approximately 3 years
Disease Control (DC) Rate | Up to approximately 3 years
Duration of Response (DoR) | Up to approximately 3 years
PFS at 6 Months | 6 months
PFS at 1 Year | 1 year
PFS at 2 Years | 2 years
OS at 6 Months | 6 months
OS at 1 Year | 1 year
OS at 2 Years | 2 years
OS at 3 Years | 3 years
Time to Progression (TTP) | Up to approximately 3 years
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to approximately 9 months
Number of Participants with TEAEs Grade 3 or Above per Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. | Up to approximately 3 years
Number of Participants with Serious TEAEs | Up to approximately 3 years
Number of Participants with TEAEs Leading to Discontinuation of Treatment | Up to approximately 3 years
Number of Participants with Fatal TEAEs | Up to approximately 3 years
Number of Participants with Treatment-related Adverse Events (AEs) | Up to approximately 9 months
Number of Participants with Adverse Events of Interest (EOI) | Up to approximately 9 months
Serum Concentrations of Tarlatamab | Day 1 up to approximately 6 months
Number of Participants with Antitarlatamab Antibody Formation | Up to approximately 9 months
Time to First Deterioration (TTD) for Physical Function as Measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 30 (EORTC-QLQ-C30) | Baseline to Week 13 and Week 25
Change in Disease Symptoms of Cough as Measured Using EORTC-QLQ LC13 | Baseline to Week 13 and Week 25
Change in Disease Symptoms of Chest Pain as Measured Using EORTC-QLQ LC13 | Baseline to Week 13 and Week 25
Change in Disease Symptoms of Dyspnea as Measured Using EORTC-QLQ LC13 | Baseline to Week 13 and Week 25
TTD for Global Health Status as Measured by EORTC-QLQ-C30 | Baseline to Week 13 and Week 25
TTD for Quality of Life as Measured by EORTC-QLQ-C30 | Baseline to Week 13 and Week 25

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (219):
- United States (37):
  - Infirmary Cancer Center, Mobile, Alabama
  - University of Southern California, Los Angeles, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Emory University, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - University of Illinois Chicago, Chicago, Illinois
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Our Lady of the Lake Cancer Institute, Baton Rouge, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Allina Health System dba Allina Health Cancer Institute, Saint Paul, Minnesota
  - Oncology Hematology Associates, Springfield, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Astera Cancer Care, East Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Montefiore Medical Center - Bronx, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Oncology Hematology Care Incorporated, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oncology Associates of Oregon, PC, Eugene, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baptist Cancer Center Memphis Thoracic, Memphis, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology - Dallas Fort Worth, Dallas, Texas
  - US Oncology Research Investigational Products Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - The Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (5):
  - Hospital Britanico de Buenos Aires, CABA, Buenos Aires
  - Instituto Alexander Fleming, Capital Federal, Buenos Aires
  - Fundacion Medica de Rio Negro y Neuquen, Cipolletti, Río Negro Province
  - Exelsus Oncologia Clinica, San Miguel de Tucumán, Tucumán Province
  - Fundacion Centro Oncológico Riojano Integral para la Investigación y Prevención del Cáncer, La Rioja
- Australia (6):
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Cancer Research South Australia, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Austria (3):
  - Medizinische Universitaet Graz, Graz
  - Universitaetsklinikum Krems, Krems
  - Landeskrankenhaus Feldkirch, Rankweil
- Belgium (9):
  - Azorg Campus Aalst - Moorselbaan, Aalst
  - Universitair Ziekenhuis Brussel, Brussels
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Ziekenhuis Oost-Limburg, Genk
  - Algemeen Ziekenhuis Maria Middelares, Ghent
  - Centres Hospitaliers Universitaires - Helora - Hopital de Mons - Site Kennedy, Mons
  - Centre Hospitalier Universitaire-Universite Catholique de Louvain Namur-Site Godinne, Yvoir
- Brazil (10):
  - Hospital Sao Rafael-Idor, Salvador, Estado de Bahia
  - Cenantron Centro Avançado de Tratamento Oncologico Ltda, Belo Horizonte, Minas Gerais
  - Santa Casa de Misericordia de Passos, Passos, Minas Gerais
  - Hospital Uopeccan, Cascavel, Paraná
  - Hospital de Clinicas de Ijui, Ijuí, Rio Grande do Sul
  - Hospital de Clinicas de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fundacao Antonio Prudente AC Camargo Cancer Center, São Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo
  - Oncoclinicas Rio de Janeiro S A, Rio de Janeiro
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - CHU de Quebec Hopital de l Enfant Jesus, Québec, Quebec
- China (31):
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Xinqiao Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The Second Attached Hospital Of Fujian Medical University, Quanzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Cangzhou Peoples Hospital, Cangzhou, Hebei
  - Jiamusi Cancer Hospital, Jiamusi, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Nanjing Chest Hospital, Nanjing, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Jiangxi Cancer hospital, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The Affiliated Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xian Jiaotong University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Peoples Hospital, Tianjin, Tianjin Municipality
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - the First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital Of Ningbo University, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
- Czechia (5):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Nemocnice Agel Ostrava-Vitkovice as, Ostrava-Vitkovice
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni nemocnice v Motole, Prague
- Denmark (3):
  - Rigshospitalet, Copenhagen
  - Regionshospitalet Godstrup, Herning
  - Odense Universitetshospital, Odense C
- France (12):
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier Regional Universitaire de Brest - Hopital Morvan, Brest
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - Centre Hospitalier - Le Mans, Le Mans
  - Centre Leon Berard, Lyon
  - Centre Hospitalier Universitaire Nord, Marseille
  - Institut regional du Cancer Montpellier, Montpellier
  - Hopital Cochin, Paris
  - Centre Hospitalier Universitaire de Nantes - Hopital Nord Laennec, Saint-Herblain
  - Centre Hospitalier Universitaire de Strasbourg - Nouvel Hopital Civil, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse - Hopital Larrey, Toulouse
  - Clinique Teissier, Valenciennes
- Germany (8):
  - Kliniken der Stadt Koeln gGmbH, Cologne
  - Universitaetsklinikum Dresden, Dresden
  - Universitaetsklinikum Essen, Essen
  - Asklepios Fachkliniken Muenchen Gauting, Gauting
  - LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Universitaetsklinikum Heidelberg, Heidelberg
  - University Hospital Muenster, Münster
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (7):
  - Henry Dunant Hospital Center, Athens
  - Sotiria General Hospital, Athens
  - Attikon University Hospital, Athens
  - Metropolitan General, Athens
  - Metropolitan Hospital, Athens
  - Saint Lukes Hospital SA, Thessaloniki
  - European Interbalkan Medical Center, Thessaloniki
- Hong Kong (2):
  - Princess Margaret Hospital, Kowloon
  - Prince of Wales Hospital, Chinese University of Hong Kong, Shatin, New Territories
- Hungary (6):
  - Semmelweis Egyetem, Budapest
  - Orszagos Koranyi Pulmonologiai Intezet, Budapest
  - Matrai Gyogyintezet, Gyöngyös
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktatokorhaz, Győr
  - Fejer Varmegyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
  - Reformatus Pulmonologiai Centrum, Törökbálint
- Beaumont Hospital, Dublin, Ireland
- Israel (4):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
- Italy (4):
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - IRCCS Istituto Oncologico Europeo, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Centro Ricerche Cliniche Di Verona Societa responsabilita limitata, Verona
- Japan (19):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi-shi, Hyōgo
  - Kanagawa Prefectural Hospital Organization Kanagawa Cancer Center, Yokohama, Kanagawa
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Okayama University Hospital, Okayama, Okayama-ken
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Saitama Medical University International Medical Center, Hidaka-shi, Saitama
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Mexico (2):
  - Health Pharma Professional Research SA de CV, Mexico City, Mexico City
  - Oncare, Mexico City, Mexico City
- Netherlands (3):
  - Universitair Medisch Centrum Groningen, Groningen
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Erasmus Medisch Centrum, Rotterdam
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii imienia Eugenii i Janusza Zeylandow, Poznan
  - Instytut Gruzlicy i Chorob Pluc, Warsaw
  - Dolnoslaskie Centrum Onkologii, Pulmonologii i Hematologii, Wroclaw
- Portugal (4):
  - Hospital da Luz, SA, Lisbon
  - Hospital Cuf Descobertas, Lisbon
  - Unidade Local de Saude de Matosinhos, EPE - Hospital Pedro Hispano, Matosinhos Municipality
  - Hospital Cuf porto, Porto
- Romania (2):
  - Institutul Oncologic Prof Dr Ion Chiricuta Cluj-Napoca, Cluj-Napoca
  - Spitalul Municipal Ploiesti, Ploieşti
- South Korea (7):
  - Chungbuk National University Hospital, Cheongju Chungbuk
  - National Cancer Center, Goyang-si Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (9):
  - Hospital Regional Universitario de Malaga, Málaga, Andalusia
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Institut Catala d Oncologia Hospitalet Hospital Duran i Reynals, L'Hospitalet de Llobregat, Catalonia
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
  - Hospital Universitario Ramon y Cajal, Madrid
- Switzerland (4):
  - Universitaetsspital Basel, Basel
  - Inselspital Bern, Bern
  - Ospedale Regionale di Bellinzona e Vali, Mendrisio
  - Kantonsspital Sankt Gallen, Sankt Gallen
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (6):
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Bagcilar Medipol Mega Universite Hastanesi, Istanbul
  - Izmir Katip Celebi Universitesi Ataturk Egitim ve Arastirma Hastanesi, Izmir
  - Medical Park Seyhan Hastanesi, Mersin
  - VM Medical Park Mersin Hastanesi, Mersin
  - Sakarya Egitim ve Arastirma Hastanesi, Sakarya

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Paulson KG, Lau SCM, Ahn MJ, Moskovitz M, Pogorzelski M, Hafliger S, Parkes A, Zhang Y, Hamidi A, Thompson CG, Wermke M. Safety and activity of tarlatamab in combination with a PD-L1 inhibitor as first-line maintenance therapy after chemo-immunotherapy in patients with extensive-stage small-cell lung cancer (DeLLphi-303): a multicentre, non-randomised, phase 1b study. Lancet Oncol. 2025 Oct;26(10):1300-1311. doi: 10.1016/S1470-2045(25)00480-2. Epub 2025 Sep 8. PMID 40934933
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com